CLINICAL TRIAL: NCT04490772
Title: Characteristics and Outcomes of Gastrointestinal Manifestations of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidi Karam, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: COVID gastro intestinal
Record Dates: First submitted 2020-07-20; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Infectious
Keywords: Covid-19; characteristics; Outcome; Egypt
MeSH Terms: conditions — Communicable Diseases; COVID-19 | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Covid-19: COVID-19 patients presented with gastrointestinal manifestations
  Interventions: Diagnostic Test: Laboratory tests

INTERVENTIONS:
Diagnostic Test: Laboratory tests — Laboratory tests such as CBC, Liver function and CRP

SUMMARY:
Patients confirmed COVID-19 with gastrointestinal manifestations will be included. Characteristics and outcomes will be described for them.

DETAILED DESCRIPTION:
Patients diagnosed as confirmed Covid-19 according to WHO and Egyptian Ministry of Health and Population (MOH) definitions will be included.The following will be done for all patients:

Demographic characters; age, sex, presence of co-morbidities such as hypretension, diabetes mellitus, obstructive lung diseases, ischemic heart diseases...etc, history of contact to covid-19 patients or recent travelling abroad.Clinical Characteristics: By recording of clinical manifestation such as fever, cough, shortness of breath, sore throat, change in taste or smell, nausea,vomiting and diarrhea will be done. Complications and the type of treatment received by the patients will also be described including mechanical ventilation.

Laboratory data will also be included : blood picture, liver enzymes, ESR,CRP, serum ferritin, D-dimer and troponin.

Follow up of the patients will be done until improvement, deaths or complications to determine disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Covid-19 with GIT manifestations

Exclusion Criteria:

* Patients refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Confirmed Covid-19 with GIT manifestations
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Clinical data questionnaire | 2 months
  Clinical characteristics of age, sex, comorbidities and symptoms.
Tests such as CBC | 2 months
  Laboratory characters
liver function test | 2 months
  Laboratory characters

IPD SHARING:
Plan to Share IPD: No